CLINICAL TRIAL: NCT04670614
Title: Regional Anesthesia (Supra-Orbital and Infra-Orbital Nerve Block) (SION) for Pain Management in Trans-sphenoidal Hypophysectomy
Acronym: SION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-15700
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Post-operative Surgical Pain
Keywords: trigeminal nerve block; trans-sphenoidal endoscopic pituitary surgery; supra-orbital nerve block; infra-orbital nerve block
MeSH Terms: interventions — Nerve Block; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve Block Procedure (Other): Supra-orbital and Infra-orbital peripheral nerve blocks with 0.5% ropivicaine
  Interventions: Procedure: Nerve Block with ropivicaine 0.5% Injectable Solution
- Placebo sham control (Sham Comparator): sham control 0.9% Normal Saline
  Interventions: Procedure: Nerve Block with Placebo sham control of 0.9% Normal Saline

INTERVENTIONS:
Procedure: Nerve Block with ropivicaine 0.5% Injectable Solution — Peripheral nerve blocks using 0.5% ropivicaine
  Arms: Nerve Block Procedure
Procedure: Nerve Block with Placebo sham control of 0.9% Normal Saline — Peripheral Nerve Block with placebo 0.9% normal saline
  Arms: Placebo sham control

SUMMARY:
This is a prospective, randomized, blinded, sham controlled regional anesthetic (supra-orbital and infra-orbital nerve block) pain study to compare the systemic postoperative pain medication requirements in patients having Trans-sphenoidal Pituitary surgery. The patients will receive general anesthesia +/- regional anesthesia for trans-sphenoidal pituitary surgery and systemic pain medication during the intra-operative and postoperative (6hrs) period. The amount of systemic pain medication requirements will be compared between those patients receiving regional and general anesthesia versus general anesthesia alone.

DETAILED DESCRIPTION:
Combined regional and general anesthesia for surgery is known to provide superior pain control in the peri-operative period (intra and post-operative). Of particular interest in neurosurgery are more rapid patient awakening and earlier ability to perform adequate post-operative neurological exam. In addition to this, regional anesthesia can decrease the total amount of systemic pain medications necessary and thus decrease their associated side effects. Consequently, less systemic pain medications can benefit the patient in many ways.

By modifying the postop pain regime to include intraoperative regional anesthesia, there could be increased patient satisfaction, and significant economic gains to the hospital through a more streamlined, shorter, more pleasant hospital course for the patient. Patients who have this trans-sphenoidal pituitary surgery are usually same day admission patients who, following their surgery, are admitted for up to 24 hours postoperatively. Usually prolonged admissions result from headache and nausea +/- vomiting. Etiology of the headache is likely multifactorial. One theory is that stimulation of the peripheral trigeminal (Cranial Nerve Number V) fibers in the V1 and V2 distribution of the face by the surgical endoscope and surgical trauma may lead to release of inflammatory mediators and post-operative migraine. It has been shown that repetitive injection of local anesthetics in the distribution of supra-orbital nerve V1 and infra-orbital nerve V2 can decrease the incidence of chronic idiopathic migraine headaches not related to surgery. By administering regional anesthesia to the patient intra-operatively during their general anesthetic for the surgery, pain scores may be reduced, PONV (postoperative nausea and vomiting) decreased, and hospital stay shortened.This study will be examining the use of regional anesthesia (infra-orbital and supra-orbital nerve blocks) combined with general anesthesia versus general anesthesia to observe the systemic opioid consumptions of adult transsphenoidal pituitary surgery patients. Secondary endpoints of the study will be: (1) presence of PONV, (2) time in PACU (post anesthesia care unit) and finally, (3) duration of hospital stay until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adult age between 18 and 65
* American Society of Anesthesiology (ASA) 1-2
* Elective pituitary tumor surgery, tumor less than or equal to 2 cm diameter within the sella and no cavernous
* sinus invasion
* Single surgeon, Dr. Kunwar
* Male and female patients
* English speaking
* Informed consent
* Not on chronic pre-opertaive pain medications (non-narcotics) in the last 1 week prior to surgery
* No opioid pain medications pre-op in the last 1 month before surgery
* No abuse of recreational drugs (cocaine, methamphetamines, THC (tetrahydrocannabinol), opioids/heroin)
* No herbal medications for pain in the 1-month prior to surgery

Exclusion Criteria:

* Age less than 18 years
* Non-English speaking
* Allergy to: Ropivicaine
* Chronic pain condition, including idiopathic migraine as defined by the ICHD (International Classification of Headache Disorders) II criteria, requiring the use of pain medications
* Inability to comprehend or adhere to study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2018-12-25 (Actual)

PRIMARY OUTCOMES:
6 hour post-operative Morphine Requirements in milligrams (mg) | 6 hours post-op
  Systemic Intravenous (IV) morphine opioid consumption in mg in 2 groups during first 6 hours post-operatively (regional + general versus only general anesthesia)

SECONDARY OUTCOMES:
Pain exposure postoperative for 6 hours | 6 hours
  Pain score out of max 10 (Scale 0-10). "O" (no Pain) and "10" (worst possible pain)
Nausea and/or vomiting for 6 hours postoperatively | 6 hours
  Nausea score out of max 10 (Scale 0-10)."O" (no nausea) and "10" (worst nausea possible). Presence of vomiting is minimum score of 5/10.
Time to discharge from Post anesthesia care unit (PACU) in minutes | post-operative period measured in minutes up to 120 minutes
  Time patient spends in PACU from entry time until discharge to the floor in minutes
Time to discharge from hospital in minutes | post-operative time up to 36 hours
  Time measured in minutes from surgery start to discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Una Srejic, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSF Moffitt Long Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srejic U, Litonius E, Gandhi S, Talke P, Maties O, Siegmueller C, Magsaysay A, Hasen D, Kunwar S, Seth R, Gibson L, Bickler P. Bilateral Superficial Trigeminal Nerve Blocks are not More Effective than a Placebo in Abolishing Post-operative Headache Pain in Pituitary Transsphenoidal Neurosurgery: A Prospective, Randomized, Doubleblinded Clinical Trial. Rev Recent Clin Trials. 2023;18(3):228-237. doi: 10.2174/1574887118666230227113217. PMID 36843368